CLINICAL TRIAL: NCT05957770
Title: Assessment of Anxiety, Depression, Sleep Quality and Quality of Life in Rheumatoid Arthritis Patients
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maha Sayed Ibrahim Abdelrahman, Principal investigator, Assiut University
Other Study IDs: 04-2023-300223
Record Dates: First submitted 2023-07-07; First posted 2023-07-24 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- cases: rheumatoid arthritis patients
- control: healthy subjects

SUMMARY:
The goal of this case control observational study is to asses anxiety, sleep, depression and quality of life in rheumatoid arthritis patients

The main aims are:

* asses anxiety, sleep, depression and quality of life in rheumatoid arthritis patients
* their relation to disease activity

we will compare rheumatoid arthritis patients to healthy subjects.

DETAILED DESCRIPTION:
All patients were subjected to clinical evaluation (full history and examination, laboratory evaluation (erythrocyte sedimentation rate [ESR], C reactive protein [CRP] and rheumatoid factor [RF]), in addition to assessment of disease activity (disease activity score in 28 joints [DAS28]-ESR

Psychological assessment was performed according to the following scales

* Hamilton Anxiety Rating Scale (HAM-A): It consists of 14 items and measures both psychic and somatic anxiety (physical complaints related to anxiety). Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where a score ≤ 17 indicates mild anxiety, 18-24 mild to moderate anxiety, , 25-30 moderate to severe anxiety and scores >30 indicate severe anxiety.
* Hamilton Depression Rating Scale: the original scale has 21 items, but scoring is based only on the first 17. Scores less than or equal to 7 indicates normal response, 8-13 mild depression, 14-18 Moderate, 19-22 severe, and > 22 very severe depression.

Sleep quality assessment was done via

* Insomnia severity index (ISI) : contains seven domains assessing sleep-onset difficulties, sleep maintenance, sleep satisfaction, effect on daily functioning, impairment attributed to sleep problems, and distress associated with insomnia. Each item is rated on a 0-4 scale, and the total score ranges from 0 to 28. A higher score suggests more severe insomnia.
* Epworth sleepiness scale : subjects describe how often they fall asleep in certain situations on a scale of 0-3, with total scores ranging from 0 to 24. An ESS score ≥ 10 is indicative of subjective excessive daytime sleepiness and score > 16 indicates high level of daytime sleepiness.

Pittsburgh Sleep Quality Index the first 4 items are open questions, whereas items 5 to 19 are rated on a 4-point Likert scale. Individual items scores yield 7 components (sleep duration, sleep disturbance, sleep latency, daytime dysfunction due to sleepiness, sleep efficiency, overall sleep quality, and sleep medication use). The scores for each component are summed to get a total score (range 0-21). A score > 5 suggests poor sleep quality.

Assessment of Health status and quality of life via short form health survey (SF36):Thirty-five of the 36 items are grouped into eight scales: physical functioning, role limitations due to physical problems, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems, and mental health. One item assesses perception of changes in health over the last year but is not used calculate scale scores. Higher scores indicate high quality of life.

ELIGIBILITY:
Inclusion criteria

• Patients diagnosed with RA according to 2010 the American College of Rheumatology (ACR)/European League Against Rheumatism classification criteria

Exclusion Criteria:

* Evidence of end-organ failures such as heart failure, a liver cell or renal failure,
* History of psychological disorders or medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with RA according to 2010 the American College of Rheumatology (ACR)/European League Against Rheumatism classification criteria.
  Healthy subjects
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of insomnia in RA patients by Insomnia severity index | 1 month
  insomnia severity index contains seven domains assessing sleep-onset difficulties, sleep
  maintenance, sleep satisfaction, effect on daily functioning, impairment attributed to sleep
  problems, and distress associated with insomnia. Each item is rated on a 0-4 scale, and th
  e total score ranges from 0 to 28. A higher score suggests more severe insomnia
evaluation of excessive daytime sleepiness by Epworth sleepiness scale | 1 month
  Subjects describe how often they fall asleep in certain situations on a scale of 0-3, with total scores ranging from 0 to 24. An ESS score ≥ 10 is indicative of subjective excessive daytime sleepiness and score > 16 indicates high level of daytime sleepiness
evaluation of anxiety in RA patients by hamilton anxiety scale | 1 month
  It consists of 14 items and measures both psychic and somatic anxiety (physical complaints related to anxiety). Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where a score ≤ 17 indicates mild anxiety, 18-24 mild to moderate anxiety, , 25-30 moderate to severe anxiety and scores >30 indicate severe anxiety
evaluation of depression in RA patients by hamilton depression scale | 1 month
  The original scale has 21 items, but scoring is based only on the first 17 with total score ranges from 0 to 52. Scores less than or equal to 7 indicates normal response, 8-13 mild depression, 14-18 Moderate, 19-22 severe, and > 22 very severe depression
evaluation of QoL in RA patients by short form health survey (sf36 ) | 1 month
  Thirty-five of the 36 items are grouped into eight scales: physical functioning, role limitations due to physical problems, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems, and mental health. One item assesses perception of changes in health over the last year but is not used calculate scale scores. Mean score ranges from 0 to100. High scores indicate lower disability.
evaluation of sleep quality and disturbances in RA patients by Pittsburgh Sleep Quality Index | 1 month
  The first 4 items are open questions, whereas items 5 to 19 are rated on a 4-point Likert scale. Individual items scores yield 7 components (sleep duration, sleep disturbance, sleep latency, daytime dysfunction due to sleepiness, sleep efficiency, overall sleep quality, and sleep medication use). The scores for each component are summed to get a total score (range 0-21). A score > 5 suggests poor sleep quality

SECONDARY OUTCOMES:
Correlation of disease activity( das28) with hamilton anxiety scale, hamilton depression scale,Epworth sleepiness scale,Pittsburgh Sleep Quality Index and short form health survey sf 36 | 1 month
  The DAS28 assessment includes a measurement of tender joint count (TJC), swollen joint count (SJC) acute phase reactant (ESR or CRP) and patient's global assessment of disease activity, which is scored from zero to 100 with higher scores indicating active disease. DAS28>5.1 indicates high disease activity. A score 3.5-5.1 indicates moderate disease activity. A score 2.6-3.2 indicates low disease activity and score <2.6 indicates remission. Score ranges from 0 to 9.4

CONTACTS AND LOCATIONS:
Overall Officials: Maha Abdelrahman, MD,PhD, Principal Investigator — Assiut University
Locations (1):
- Faculty of medicine, Assiut university hospital, Asyut, Egypt